CLINICAL TRIAL: NCT07405736
Title: Lubiprostone Combined With Maintenance Therapy for Prevention of Postoperative Recurrence in Peritoneal Metastatic Colorectal Cancer, A Randomized Controlled Phase II Study
Brief Title: Lubiprostone Combined With Maintenance Therapy for Prevention of Postoperative Recurrence in Peritoneal Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Director, Department of Colorectal Surgery; Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-439
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer Metastatic; Peritoneal (Metastatic) Cancer; Peritoneal Metastasis; Colorectal Cancer (CRC); MSS Metastatic Colorectal Cancer
Keywords: Peritoneal metastasis; Colorectal cancer; Maintenance therapy; Lubiprostone; Cytoreductive Surgery; Progression-free survival
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Colorectal Neoplasms | interventions — Maintenance; Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigator-Selected Maintenance Therapy + Lubiprostone (Experimental): Participants receive investigator-selected standard-of-care maintenance therapy plus lubiprostone (24 μg orally twice daily) during the maintenance period, until disease progression, unacceptable toxicity, withdrawal, or other protocol-defined discontinuation criteria.
  Interventions: Drug: maintenance therapy plus lubiprostone
- Investigator-Selected Maintenance Therapy (Active Comparator): Participants receive investigator-selected standard-of-care maintenance therapy during the maintenance period, until disease progression, unacceptable toxicity, withdrawal, or other protocol-defined discontinuation criteria.
  Interventions: Drug: maintenance therapy

INTERVENTIONS:
Drug: maintenance therapy plus lubiprostone — In experiment arm, participants receive investigator-selected standard-of-care maintenance therapy plus lubiprostone (24 μg orally twice daily) during the maintenance period, until disease progression, unacceptable toxicity, withdrawal, or other protocol-defined discontinuation criteria.
  Arms: Investigator-Selected Maintenance Therapy + Lubiprostone
Drug: maintenance therapy — In active comparator arm, participants receive investigator-selected standard-of-care maintenance therapy during the maintenance period, until disease progression, unacceptable toxicity, withdrawal, or other protocol-defined discontinuation criteria.
  Arms: Investigator-Selected Maintenance Therapy

SUMMARY:
The goal of this phase II randomized controlled clinical trial is to evaluate whether adding lubiprostone to standard postoperative maintenance therapy can delay disease progression and recurrence in adult patients with colorectal cancer and peritoneal metastases (PM-CRC) who have undergone cytoreductive surgery with or without HIPEC after systemic treatment. The main questions it aims to answer are:

Does lubiprostone plus maintenance therapy improve the 1-year progression-free survival (PFS) rate compared with maintenance therapy alone?

Is lubiprostone safe and feasible for long-term use during the maintenance period in this PM-CRC population?

Researchers will compare lubiprostone + maintenance therapy versus maintenance therapy alone to see if the addition of lubiprostone prolongs PFS, reduces the risk of distant metastasis, improves overall survival, and maintains or improves quality of life.

Participants will:

Be randomly assigned to receive maintenance therapy with lubiprostone or maintenance therapy alone after surgery (CRS ± HIPEC) and prior systemic therapy, according to the study protocol.

Undergo scheduled follow-up assessments for disease status (progression/recurrence), survival outcomes, treatment-related toxicity, and quality of life using the EORTC QLQ-C30 (v3.0) questionnaire.

DETAILED DESCRIPTION:
Peritoneal metastasis (PM) is a distinct and clinically challenging dissemination pattern of colorectal cancer (CRC), often associated with limited intraperitoneal drug penetration, fibrotic remodeling, and an immunosuppressive peritoneal microenvironment. Despite intensive multimodal treatment-including systemic therapy and cytoreductive surgery (CRS) with or without hyperthermic intraperitoneal chemotherapy (HIPEC)-postoperative recurrence and progression remain common, and the role of postoperative maintenance strategies in PM-CRC is not well established.

Preclinical work conducted by the study team supports a role for purinergic signaling, particularly the P2Y receptor axis (e.g., P2RY2), in processes relevant to peritoneal implantation and stromal remodeling. In these models, lubiprostone demonstrated inhibitory effects on P2RY2-associated signaling and showed peritoneum-focused antitumor activity when combined with systemic chemotherapy, with a favorable tolerability profile at treatment-relevant exposures. Together, these observations provide the scientific rationale to evaluate lubiprostone as a low-toxicity, accessible candidate for long-term postoperative maintenance to delay recurrence or progression in patients with CRC and peritoneal metastases who have undergone adequate cytoreduction.

This study is a prospective, open-label, randomized, controlled phase II trial. Participants will be randomized 1:1 to receive either investigator-selected standard-of-care (SOC) maintenance therapy alone or SOC maintenance therapy plus lubiprostone. Randomization will use a block allocation sequence generated by an independent statistician. Because the study compares a pharmacologic add-on strategy to SOC maintenance, blinding is not applied.

SOC maintenance therapy is individualized by treating investigators according to contemporary guideline-based practice and patient-specific factors (e.g., prior systemic therapy exposure, performance status, age, molecular profile, and primary tumor location). The protocol specifies permitted maintenance approaches and rules for regimen selection and modification; however, the study does not mandate a single uniform maintenance regimen across all participants. Lubiprostone is administered orally during the maintenance period, and treatment may continue until protocol-defined discontinuation criteria are met (e.g., disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-specified reasons). The protocol includes guidance for temporary interruption or dose adjustment of lubiprostone to manage treatment-emergent adverse events.

Disease status is evaluated using standardized imaging procedures to ensure consistency across participants. Cross-sectional imaging is performed at protocol-defined intervals; when conventional imaging is indeterminate, ^68Ga-FAPI PET/CT may be used to clarify disease status per protocol guidance and local availability. Tumor burden and peritoneal disease distribution may be documented using a standardized regional approach, including peritoneal cancer index (PCI) assessment performed according to the protocol workflow (e.g., independent radiology review).

Safety surveillance includes routine clinical assessments and laboratory monitoring during study treatment and for a defined period after the last study-related treatment. Adverse events are collected systematically, graded using standard toxicity criteria specified in the protocol, and reported according to applicable regulatory and oversight requirements. The protocol highlights management considerations for anticipated lubiprostone-associated gastrointestinal symptoms (e.g., nausea, diarrhea, abdominal discomfort) and emphasizes prompt evaluation for suspected mechanical gastrointestinal obstruction.

The statistical analysis plan evaluates whether adding lubiprostone to SOC maintenance shows a superiority signal on time-to-event efficacy outcomes, with primary analyses conducted in the intention-to-treat population and supportive analyses in the per-protocol population. Safety analyses include participants who receive at least one dose of study-related treatment as defined in the protocol. No interim efficacy analysis is planned; ongoing safety data are reviewed through an independent safety monitoring process.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participates and provides written informed consent.
* Histologically confirmed colon/rectal adenocarcinoma with molecular status confirmed as pMMR or MSS.
* Cytoreductive surgery (CRS) achieves CC0/CC1 cytoreduction.
* No extraperitoneal metastasis prior to treatment.
* ECOG performance status 0-1 with adequate organ function per protocol requirements.

Exclusion Criteria:

* Extensive multisystem metastases on baseline imaging assessment.
* Tumor carrying BRAF V600E mutation.
* dMMR/MSI-H, or confirmed pathogenic POLE/POLD1 mutation(s).
* Cachexia or decompensated organ dysfunction.
* History of another malignancy within the past 5 years.
* Known or suspected hypersensitivity/allergy to the study drug or related formulations.
* Multiple primary cancers.
* Any serious disease or other medical, psychological, or social condition that, in the investigator's judgment, may compromise participant safety or affect study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
1-year Progression-Free Survival (PFS) Rate | From randomization to 12 months (1 year).
  Progression-free survival is defined as the time from randomization to the first documented recurrence/progression event. Recurrence/progression is confirmed by at least one of the following:
  imaging assessment judged as recurrence by two radiologists; or physical examination + progressively rising tumor markers and/or MRD and other objective evidence supporting progression; or positive cytology/histology from biopsy.
  The date of recurrence is the date the above diagnostic confirmation is established; isolated CEA rise alone is not sufficient evidence of recurrence.

SECONDARY OUTCOMES:
3-year Progression-Free Survival (PFS) rate | From randomization to 36 months (3 years).
  PFS is defined as the time from randomization to the first documented recurrence/progression event, using the same event confirmation rules as above (radiology/clinical objective evidence/positive pathology). Tumor assessments are performed at scheduled intervals (every 3 months or 6 months) and/or whenever clinical signs suggest progression.
3-year Overall Survival (OS) Rate | From randomization to 36 months (3 years).
  Overall survival is defined as the time from randomization to death from any cause. Participants alive at the last follow-up are censored on that date.
Extraperitoneal (Distant) Metastasis Rate | Up to 36 months (3 years) after randomization.
  Proportion of participants who develop metastasis outside the peritoneum (extraperitoneal organs/tissues) during follow-up, confirmed by imaging and/or pathology.
Treatment Toxicity (Adverse Events) | From start of study treatment through 30 days after the end of treatment.
  Treatment-emergent adverse events graded and recorded according to NCI CTCAE v5.0, with emphasis on the incidence of Grade ≥3 adverse events.
Quality of Life Evaluated by EORTC QLQ-C30 v3.0 | Baseline; every 3 months during treatment; and at end of follow-up (up to 36 months).
  Quality of life assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30), version 3.0. Scores are linearly transformed to 0-100 scales. For the Global Health Status/QoL scale, higher scores indicate better quality of life. For Functional Scales (physical, role, emotional, cognitive, social), higher scores indicate better functioning. For Symptom Scales/Items (fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties), higher scores indicate worse symptom burden/problems. The questionnaire is administered at baseline, every 3 months during treatment, and at the end of follow-up to compare longitudinal QoL differences between treatment groups.

IPD SHARING:
Plan to Share IPD: No